CLINICAL TRIAL: NCT04225299
Title: An Evaluation of the Efficacy of Partial Gland Ablation (PGA) With TOOKAD® Vascular Targeted Photodynamic Therapy (VTP) Versus Active Surveillance for Men With Intermediate Risk Localized Prostate Cancer
Brief Title: Evaluation of Efficacy of TOOKAD® (VTP) Versus Active Surveillance for Intermediate Risk Localized Prostate Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA didn't approve the design of the protocol so we didn't start the study
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1901 PCM306
Record Dates: First submitted 2019-12-26; First posted 2020-01-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Localized Prostate Cancer
Keywords: Prostatic Disease; Genital Neoplasm,male; Urogenital neoplasm; Genital disease,male; Male urogenital disease; Neoplasms; Neoplasms by site; Prostatic neoplasm; Carcinoma
MeSH Terms: conditions — Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Prostatic Neoplasms; Carcinoma | interventions — palladium-bacteriopheophorbide; padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TOOKAD® (Experimental): TOOKAD® , lyophilized formulation, given at a dose of 4mg/Kg.
  Interventions: Drug: TOOKAD®
- Active Surveillance (No Intervention): Active surveillance is one of the management strategy in men who have intermediate risk localised prostate cancer

INTERVENTIONS:
Drug: TOOKAD® — TOOKAD® -VTP procedure will consist of an IntraVenous (IV) administration to patients using a 753nm laser light at a fixed power of 150mW/cm and a fixed energy at 200J/cm delivered through transperineal interstitial optical fibers. The needles are positioned in the prostate under ultra sound image guidance
  Other Names: WST11
  Arms: TOOKAD®

SUMMARY:
Multi-center, prospective, randomized controlled clinical trial that will compare two treatment methods (PGA with TOOKAD® VTP and Active Surveillance) for treating localized prostate cancer. The study will include criteria for evaluation, biopsy, eligibility, informed consent, subsequent management and decision making conducted based on data provided locally at each center that follow a set of standardized criteria.

DETAILED DESCRIPTION:
The primary endpoint requires follow-up through 30 months, but all subjects will be followed for 72 months regardless of initiation of other local or systemic prostate cancer treatments, which will allow assessments of recurrence rates and morbidity after conversion to radical therapy, long-term safety and tolerability, as well as oncologic outcomes.

This is multi-center, prospective, randomized controlled phase III clinical trial that will compare two treatment methods (PGA with TOOKAD® VTP and Active Surveillance) for treating localized prostate cancer who meet the inclusion criteria will be approached for participation in the clinical study. Patients consenting to participate will be individually randomized to TOOKAD® VTP or Active Surveillance with a 1:1 ratio. Central randomization will be performed using an independent web-based allocation system. Randomization will be stratified by center using minimization. Ongoing assessment of patients in both arms will be balanced, including follow up examinations, PSA testing, MRI and biopsies at defined intervals.

Subjects in the experimental arm will receive the experimental treatment consisting of unilateral TOOKAD® VTP treatment applied to the index lobe containing pattern 4 cancer. The treatment will be administered under general anesthesia. Routine ultrasound examination in the operating room will be performed for morphometric description of the prostate and to facilitate accurate treatment planning and probe placement. Ultrasound will not be used for diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 years or older.
2. Men who have chosen Active Surveillance as the treatment for their prostate cancer.
3. Patients who have had a multiparametric MRI of the prostate performed and have undergone transrectal systematic biopsy plus biopsy of any lesions (or "areas") considered suspicious per the MRI (PIRADS version 2 score of 4 or 5) within 6 months before signing consent.
4. Unilateral Grade Group 2 (Gleason grade 3+4=7) prostate cancer with a total length of Gleason pattern 4 no more than 2mm when measured in all systematic biopsy cores plus up to 1 core from each targeted biopsy lesion (if more than 1 core is taken from a given lesion the core with the longest length of pattern 4 will be included). Note: the presence and length of Grade Group 1 (Gleason score 3+3=6) cancer in the biopsy will not be considered when determining eligibility.
5. Prostate cancer clinical stage up to cT2a, N0/Nx, M0/Mx.
6. Prostate volume ≥20 mL and ≤80 mL
7. Serum PSA ≤10 ng/mL.
8. Patients with cT2a and PSA between 10 and 20 ng/mL will have appropriate imaging and work up to sufficiently exclude clinical evidence of bone metastases (e.g., bone scan, whole body MRI, PET scan, or equivalent). Patients with sites considered "suspicious" may be evaluated with confirmatory biopsy to determine eligibility. Patients with sites considered "definite" or "consistent with" bone metastases will be excluded.
9. Men who are sexually active with women of childbearing potential must use contraceptive method with a failure rate of less than 1% per year. Contraception should be continued for a period of 90 days after the VTP procedure. The individual methods of contraception may be determined in consultation with the investigator.
10. Signed Informed Consent Form.

Exclusion Criteria:

1. Grade Group 3, 4 or 5 (≥ Gleason Score 4+3=7) cancer
2. In patients with Grade Group 2 cancers, a total length of Gleason pattern 4 more than 2mm when measured in all systematic biopsy cores plus up to 1 core from each targeted biopsy lesion (if more than 1 core is taken from a given lesion, include the mm of pattern 4 in the 1 core with the longest length of pattern 4)
3. Bilateral GG 2 cancer
4. MRI evidence of extracapsular extension of cancer (MRI read as "definite", "frank" or "gross" ECE, or MRI lesion with >10mm capsular contact, in an area with biopsy proven cancer).
5. Seminal vesicle invasion on DRE or MRI ("probable" or "consistent with")
6. Radiographically suspicious lymph node involvement confirmed with biopsy or PET scan.
7. Any prior or current treatment for prostate cancer, including but not limited to surgery, radiation therapy (external or brachytherapy) or chemotherapy;
8. Life expectancy less than 10 years;
9. Participation in another clinical study involving an investigational product that in the opinion of the investigator may interfere with the endpoints or investigational criteria of this study;
10. Inability to understand the informed consent document, to give consent voluntarily or to complete the study tasks, especially inability to understand and fulfill the health-related QOL questionnaire;
11. Any history of a definitively ablative procedure for benign prostatic disease, such as benign prostatic hyperplasia, including TURP, whether electrosurgical or thermal laser ablation; or high intensity frequency ultrasound (HIFU) or cryotherapy, for focal or total ablative therapy of the prostate.
12. Any condition or history of illness or surgery that may pose an additional risk to men undergoing the VTP procedure such as:

    1. Medical conditions that preclude the use of general anesthesia;
    2. Any condition or history of active rectal inflammatory bowel disease or other factors which might increase the risk of fistula formation;
    3. Hormonal manipulation (excluding 5-alpha-reductase inhibitors) that alters androgen production within the previous 6 months;
    4. Oral anticoagulant drugs that could not be withdrawn at least 5 days prior to the VTP procedure or antiplatelet drugs (e.g. aspirin) that could not be withdrawn at least 5 days prior to the VTP procedure and for at least 3 days after VTP;
    5. Renal and hepatic disorders with values of >1.5 times the upper limit of normal (ULN) or blood disorders (upon clinician judgment);
    6. A history of sun hypersensitivity or photosensitive dermatitis.
    7. Any other condition or history of illness or surgery that in the opinion of the investigator might affect the conduct and results of the study or pose additional risks to the patient (e.g., cardiac or respiratory disease precluding general anesthesia, active urethral stricture disease).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-31 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of objective progression | over 30 months
  To evaluate the difference in the rate of objective progression of cancer between men treated with TOOKAD -VTP and men managed with Active Surveillance for localized prostate cancer.

SECONDARY OUTCOMES:
Rate of conversion to radical local or systemic therapy | over 30 and 72 months
  To confirm the differences between men treated with VTP and men managed with Active Surveillance in overall rate of conversion to radical local or systemic therapy
Rate of conversion to radical local or systemic therapy following objective progression | over 30 and 72 months
  To confirm the differences between men treated with VTP and men managed with Active Surveillance in overall rate of conversion to radical local or systemic therapy following objective progression
Rate of biopsy progression in the index lobe | at 30 and 72 months
  To confirm the differences between men treated with VTP and men managed with Active Surveillance in the rate of biopsy progression in the index lobe (the lobe initially diagnosed with GG2 cancer) defined as:
  * Any Grade Group 3 or higher cancer in a biopsy core of the index lobe
  * Increase in total length of Gleason pattern 4 >1mm above baseline and >2mm in total length in a follow-up biopsy of the index lobe
Rate of clinical local or distant progression | Screening,Month 12, Month 24,Month 42 and Month 60
  The rate of clinical local or distant progression defined as any of the following:
  * Clinical stage ≥ T3N0M0 cancer
  * MRI evidence of extracapsular extension of cancer (MRI read as "definite", "frank" or "gross" ECE, or MRI lesion with >10mm capsular contact) in an area with biopsy proven cancer.
  * Seminal vesicle invasion, identified as "probable" or "definite," on DRE or MRI
  * Radiographically suspicious lymph node involvement confirmed with biopsy or PET scan.
  * Metastatic disease
  * Prostate cancer-specific death
Adverse events and Serious Adverse events | Screening-Month 72
  The rate, severity, onset and duration of adverse events (AEs) and serious adverse events (SAEs)
FACT-P - Question GP5 - Bother Related to Adverse Events | Screening,Week 2, Week 4, Week 6, Week 8, Month 3, Month 4, Month 5, Month 6, Month 12, Month 18, Month 24, and Month 36
  The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being. Only Question GP5 will be assessed to determine bother related to adverse events.
Urinary:PRO-CTCAE - Urinary Questions 61 - 65 | Screening,Week 2, Week 4, Week 6, Week 8, Month 3, Month 4, Month 5, Month 6, Month 12, Month 18, Month 24, and Month 36
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a new patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities. These include symptomatic toxicities such as pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient perspective. Only Urinary Questions 61 - 65 will be assessed
Pain: PRO-CTCAE Pain Question 48 | Screening,Week 2, Week 4, Week 6, Week 8, Month 3, Month 4, Month 5, Month 6, Month 12, Month 18, Month 24, and Month 36
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a new patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities. These include symptomatic toxicities such as pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient perspective.Only Pain Question 48 will be assessed
Bowel Symptoms: PRO-CTCAE questions 17 and 18 | Screening,Week 4, Week 8, Month 3, Month 6, Month 12, Month 18, Month 24, and Month 36, Month 48, Month 60, and Month 72
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a new patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities. These include symptomatic toxicities such as pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient perspective. Only Bowel Symptoms questions 17 and 18 will be assessed
Sexual Function: PRO-CTCAE questions 66-68 and 70-72 | Screening,Week 4, Week 8, Month 3, Month 6, Month 12, Month 18, Month 24, and Month 36, Month 48, Month 60, and Month 72
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a new patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities. These include symptomatic toxicities such as pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient perspective. Only Sexual Function questions 66-68 and 70-72 will be assessed
Anxiety = PRO-CTCAE question 54 | Screening,Week 4, Week 8, Month 3, Month 6, Month 12, Month 18, Month 24, and Month 36, Month 48, Month 60, and Month 72
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a new patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities. These include symptomatic toxicities such as pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient perspective.Only Anxiety question 54 will be assessed
Anxiety = MAX-PC Questions 15-18 - Anxiety related to fear of prostate cancer recurrence | Screening,Month 6, Month 12, Month 18, Month 24, and Month 36, Month 48, Month 60, and Month 72
  The Memorial Anxiety Scale for Prostate Cancer (MAX-PC) has been developped to facilitate the identification and assessment of men with prostate cancer-related anxiety. This scale consists of three subscales that measure general prostate cancer anxiety, anxiety related to prostate specific antigen (PSA) levels in particular, and fear of recurrence. Only Anxiety Questions 15-18 will be assessed
Assessment feasibility of performing radical, local or systemic treatment | within 90 days after treatment
  The physician will evaluate the ease or difficulties of radical, local or systemic therapy after VTP procedure using a scale . The instrument to be used to assess feasibility of performing RT will be a 5-point Likert Scale.
  The question may be similar to the following:
  "What was the difficulty in performing radical treatment on the subject" and proposed anwers will be: None, Minimal, Moderate, Severe or Extreme
Safety of radical, local or systemic treatment | within 90 days after treatment
  Safety recorded as incidence of Adverse events and Serious Adverse Events
Biochemical outcomes of radical, local or systemic treatment | 6 weeks and 24 months after treatment
  Biochemical Response recorded as serum PSA change as absolute measurement in ng/dL and as percentage increase or decrease over time
Clinical recurrence | 6 weeks and 24 months after treatment
  Clinical recurrence recorded as physician recorded objective recurrence of tumor on physical exam or imaging.
Primary cause for conversion to radical treatment | Over 30 and 72 months
  Identification of the primary cause for conversion to radical treatment as assessed by physician:
  * Pre-defined cancer progression
  * Changes in clinical parameters in absence of objective progression (physicial examination findings, PSA, imaging (MRI, CT, PET), biopsy, or other tests to be documented such as genomic tests)
  * Significant change in anxiety about prostate cancer (Defined as increase of last MAX-PC (Memorial Anxiety Scale for Prostate Cancer)-fear of recurrence score prior to conversion to radical therapy by 3 points or more vs. baseline) in the absence of objective progression or change in clinical parameters
  * Patient preference in absence of objective progression, change in clinical parameters, or documented prostate cancer anxiety
Assessment of PSA Level | Screening, Day of VTP ,Month 6, Month 18, Month 30, Month 36, Month 48 and Month 72
  Assessment of PSA level in predicting or monitoring oncologic outcomes of local recurrence, and local or systemic progression. PSA serum level to be recorded as ng/ml
Assessment of PSA density | Screening, Day of VTP ,Month 6, Month 18, Month 30, Month 36, Month 48 and Month 72
  Assessment of PSA density in predicting or monitoring oncologic outcomes of local recurrence, and local or systemic progression. PSA density is calculated as total PSA (ng/ml) divided by prostate volume (ml).
Assessment of PSA kinetics | Screening, Day of VTP ,Month 6, Month 18, Month 30, Month 36, Month 48 and Month 72
  Assessment of PSA kinetics in predicting or monitoring oncologic outcomes of local recurrence, and local or systemic progression. PSA kinetics is evaluated as change in PSA serum level in ng/ml over time.
Assessment of MRI dynamic characteristics (change in size of initial lesions) | Screening, Month 12,Month 24, Month 42 and Month 60
  Change in size of initial lesion on MRI in cm3
Assessment of MRI dynamic characteristics (change in PIRADS v2 score of initial lesions) | Screening, Month 12,Month 24, Month 42 and Month 60
  Change in PIRADS v2 Score of initial lesion
Assessment of MRI dynamic characteristics (Development of new lesions) | Month 12,Month 24, Month 42 and Month 60
  Incidence of new lesions discovered
Assessment of MRI dynamic characteristics (Changes in level of suspicion for ECE, SVI, LN metastases) | Screening, Month 12,Month 24, Month 42 and Month 60
  Changes in imaging results to indicate potential progression of prostate cancer outside the prostate gland (Changes in level of suspicion for Extra Capsular Extension (ECE), Semical vesicle invasion (SVI), Lymph node (LN) metastases used to identify local recurrence, and local, regional or distant progression).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coleman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States